CLINICAL TRIAL: NCT02587104
Title: A Single Center, Prospective, Non-Randomized, Historical Controlled Trial of dHACM In the Treatment of Diabetic Foot Ulcers
Brief Title: dHACM In the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFDFU009
Record Dates: First submitted 2015-09-25; First posted 2015-10-27 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetes Mellitus; Foot Diseases; Foot Ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Diseases; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EpiFix (Experimental): Weekly application of EpiFix and standard of care (moist wound therapy and offloading)
  Interventions: Other: EpiFix

INTERVENTIONS:
Other: EpiFix — Weekly application of EpiFix and standard of care (moist wound therapy and offloading)

SUMMARY:
A single-centered, non-randomized study with approximately 20 subjects that will be seen for up to 12 weeks, each receiving the EpiFix plus standard of care. Safety and effectiveness will be monitored throughout the study.

DETAILED DESCRIPTION:
Approximately 20 subjects will be enrolled in this study. Subjects will be seen for up to12 weeks unless 100% epithelialization of the index wound and two subsequent healing confirmation visits have been achieved prior to week 12. Each subject will receive a weekly application of the EpiFix plus standard of care until 100% epithelialization is achieved. The subjects will be evaluated for efficacy and safety during the course of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with a DFU that meets all of the following requirements:

   * Wound diabetic in origin
   * Located on the dorsal or plantar surface of the foot
   * Size ranging from 1 to 25 cm2 (Debridement will be done prior to measurement and treatment, if clinically indicated)
   * Open a minimum of 30 days prior to treatment (Day 0)
   * Failure of prior treatment to heal the wound (≤25% wound area reduction after 14 consecutive days of offloading and moist wound therapy immediately prior to treatment on Day 0)
2. Affected limb must demonstrate adequate circulation, as demonstrated by one of the tests listed below (completed <60 days prior to Day 0)

   * Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg; or
   * ABIs with results of ≥0.7 and ≤1.2; or
   * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected foot
3. General Subject Characteristics:

   * Age 18 or older
   * Type 1 or 2 Diabetic (criteria for the diagnosis of diabetes mellitus per ADA)
   * Willing and able to provide consent and participate in all procedures necessary to complete the study
   * Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence)

Exclusion Criteria:

1. DFUs meeting any of the criteria below:

   * Non-Index wounds within 2 cm of the index DFU
   * Active infection at index DFU
   * Index DFU greater than one year in duration without intermittent closure
   * DFU is a possible non-revascularizable surgical site
   * Known or suspected local skin malignancy to the index diabetic ulcer
   * Index DFU treated with biomedical or topical growth factor within the previous 30 days. Study ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®), EpiFix®, or other scaffold materials (e.g. Oasis®, MatriStem®) within the last 30 days
2. Subjects with the following lab values at Day 0:

   * HbA1C ≥ 12% at any time within previous 60 days
   * Serum Creatinine ≥ 3.0mg/dl within last 6 months
3. Therapy Related Exclusions:

   * Subjects previously or currently enrolled in this study
   * Subjects being treated with investigational drug(s) or investigational therapeutic device(s) within 30 days
   * Subjects currently receiving radiation therapy or chemotherapy
   * Currently being treated with antibiotics
4. Other Exclusion Criteria:

   * Active Charcot deformity or major structural abnormalities of the foot
   * Known allergy to Gentamicin sulfate or Streptomycin sulfate
   * Subjects diagnosed with autoimmune connective tissue diseases
   * Any pathology that would limit the blood supply and compromise healing
   * Known history of poor compliance with medical treatments
   * Subjects who are known to be pregnant, plan to become pregnant, or are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with complete closure of the study ulcer | 12 weeks
  The percentage of subjects with complete closure of the study ulcer as assessed by photographic evaluation
The proportion of product related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events | 12 weeks
  The proportion of product related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events at 12 weeks.

SECONDARY OUTCOMES:
Time to complete closure | up to 12 weeks
  As assessed by photographic evaluation and the Investigator
Rate of wound closure | up to 12 weeks
  As assessed by photographic evaluation and the Investigator
Incidence of ulcer recurrence | up to 12 weeks
  Incidence of ulcer recurrence at the site of the study ulcer
Quality of Life -Health Survey | up to 12 weeks
  Change in quality of life metrics as measured by SF-36 Health Survey
Quality of Life- Pain Score | up to 12 weeks
  Changes in the patients reported pain scores as measure by the Visual Analog Scale
Cost effectiveness of treatment of dHACM | up to 12 weeks
  Measuring the amount of product usage

CONTACTS AND LOCATIONS:
Overall Officials: Perry Mayer, MD, Principal Investigator — The Mayer Institute
Locations (1):
- The Mayer Institute, Hamilton, Ontario, Canada